CLINICAL TRIAL: NCT04682353
Title: A Randomized, Dose-range Finding Study to Evaluate Pharmacokinetics of Medroxyprogesterone Acetate Following a Single Subcutaneous Administration of TV-46046 in Healthy Women of Reproductive Age
Brief Title: A Study to Evaluate the Pharmacokinetics (PK) of Medroxyprogesterone Acetate Following an Injection of TV-46046 in Healthy Women of Reproductive Age
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Collaborators: FHI 360 (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: TV46046-WH-10159
Record Dates: First submitted 2020-12-04; First posted 2020-12-23 (Actual); Results first posted 2024-02-26 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2023-07

CONDITIONS: Contraception
Keywords: Pharmacokinetics
MeSH Terms: interventions — Medroxyprogesterone Acetate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group 1 - 120 mg/0.4 mL (Experimental)
  Interventions: Drug: TV-46046
- Group 2 - 180 mg/0.6 mL (Experimental)
  Interventions: Drug: TV-46046
- Group 3 - 240 mg/0.8 mL (Experimental)
  Interventions: Drug: TV-46046
- Group 4 - 104 mg/0.65 mL (Active Comparator)
  Interventions: Drug: Depo-subQ Provera

INTERVENTIONS:
Drug: TV-46046 — SC injection of 300 mg/mL (120 mg/0.4mL; 180 mg/0.6mL; 240 mg/0.8mL)
  Arms: Group 1 - 120 mg/0.4 mL; Group 2 - 180 mg/0.6 mL; Group 3 - 240 mg/0.8 mL
Drug: Depo-subQ Provera — SC injection of 104 mg/0.65 mL
  Arms: Group 4 - 104 mg/0.65 mL

SUMMARY:
The primary objective of this study is to evaluate and compare the pharmacokinetic profile of Medroxyprogesterone acetate following subcutaneous administration of 3 different doses of TV-46046 and a dose of Depo-subQ Provera in healthy female participants.

The secondary objectives of the study are to evaluate and compare the safety, local tolerability, and acceptability of a subcutaneous injection of 3 different doses of TV-46046 and a dose of Depo-subQ Provera in healthy female participants.

The total duration of the study for each participant is expected to be up to 19.5 months.

ELIGIBILITY:
Inclusion Criteria:

* has regular menstrual cycle (21 to 35 days)
* has a low risk of pregnancy (ie, sterilized, in exclusively same-sex partnership, abstinent, in monogamous relationship with vasectomized partner, using nonhormonal intrauterine device (IUD), or consistently using barrier methods of contraception)
* had a normal mammogram within the last year, if 40 years of age or older

NOTE- Additional criteria apply, please contact the investigator for more information.

Exclusion Criteria:

* has multiple risk factors for cardiovascular disease (eg, smoking, obesity, hypertension, known low HDL, high LDL, or high triglyceride levels)
* has current or history of ischemic heart disease
* has active thrombophlebitis, current or past history of thromboembolic disorders, cerebral vascular disease or stroke
* has systemic lupus erythematosus
* has rheumatoid arthritis on immunosuppressive therapy
* has unexplained vaginal bleeding
* has diabetes
* has strong family history of breast cancer (defined as one or more first degree relatives with breast cancer, breast cancer occurring before menopause in three or more family members, regardless of degree of relationship, and any male family member with breast cancer)
* has current or history of breast cancer, or undiagnosed mass detected by breast exam
* has current or history of cervical cancer
* has cirrhosis or liver tumors
* has known osteoporosis or osteopenia
* has history of diagnosed clinical depression or bipolar disorder, with or without suicidal ideation, and/or history of suicide attempt, except short-lived situational depression that did not require medication and has not recurred in last five years
* used MPA-containing injectable products in the past 12 months
* used a combined injectable contraceptive in the past 6 months
* used any of the following medications within 1 month prior to enrollment:
* any investigational drug
* oral contraceptives, contraceptive ring or patch
* levonorgestrel intrauterine system (LNG IUS) or contraceptive implant
* is participating in another clinical trial
* is pregnant
* desires to become pregnant in subsequent 24 months
* has been pregnant in last 3 months
* is currently lactating

NOTE- Additional criteria apply, please contact the investigator for more information.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2020-12-14 (Actual); Primary Completion 2022-07-11 (Actual); Study Completion 2023-01-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teva Medical Expert, MD, Study Director — Teva Branded Pharmaceutical Products R&D, Inc.
Locations (3):
- United States (2):
  - Teva Investigational Site 14002, Cypress, California
  - Teva Investigational Site 14003, San Antonio, Texas
- Teva Investigational Site 18001, Santo Domingo, Dominican Republic

IPD SHARING:
Plan to Share IPD: Yes
Upon primary clinical trial manuscript publication, researchers may request access to underlying study data. Each accepted article must be accompanied by a Data Availability Statement that describes where any primary data, associated metadata, original software, and any additional relevant materials necessary to understand, assess, and replicate the reported study findings in totality can be found. Underlying study data will be de-identified and study documents will be redacted to protect the privacy of trial participants and to protect commercially confidential information. Requests will be reviewed for scientific merit, product approval status, and conflicts of interest. Please email manuscript primary author to make your request.

RESULTS

PARTICIPANT FLOW:
Groups:
- TV46046 Dose A: Participants received a single subcutaneous (SC) injection of TV-46046 Dose A.
- TV46046 Dose B: Participants received a single SC injection of TV-46046 Dose B.
- TV46046 Dose C: Participants received a single SC injection of TV-46046 Dose C.
- Depo-subQ Provera: Participants received a single SC injection of Depo-subQ Provera.
Period: Overall Study
Arm/Group | TV46046 Dose A | TV46046 Dose B | TV46046 Dose C | Depo-subQ Provera
Started | 16 | 15 | 14 | 15
Received at Least 1 Dose of Study Drug | 16 | 15 | 14 | 15
Completed | 16 | 13 | 14 | 14
Not Completed | 0 | 2 | 0 | 1
Not completed — Lost to Follow-up | 0 | 1 | 0 | 1
Not completed — Personal reasons | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all randomized participants who received an injection of study drug.
Groups:
- TV46046 Dose A: Participants received a single SC injection of TV-46046 Dose A.
- Total: Total of all reporting groups
Arm/Group | TV46046 Dose A | TV46046 Dose B | TV46046 Dose C | Depo-subQ Provera | Total
Number analyzed (Participants) | 16 | 15 | 14 | 15 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.3 (6.1) | 33.9 (7.2) | 31.2 (7.2) | 32.9 (6.3) | 33.4 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 15 | 14 | 15 | 60
  Male | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 4 | 1 | 5 | 11
  White | 8 | 4 | 5 | 4 | 21
  More than one race | 7 | 7 | 7 | 6 | 27
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Serum Concentration (Cmax) of Medroxyprogesterone Acetate (MPA)
Time Frame: Day 0 to Day 365
Population: Pharmacokinetic (PK) analysis set included all randomized participants who received an injection of study drug, excluding any participants who had a baseline MPA concentration that exceeded 5% of their individual Cmax, had an important protocol deviation that may affect interpretation of their MPA data, or failed to provide at least 1 evaluable post-treatment MPA specimen.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms (ng)/ milliliter (mL)
Arm/Group | TV46046 Dose A | TV46046 Dose B | TV46046 Dose C | Depo-subQ Provera
Number analyzed (Participants) | 16 | 15 | 14 | 14
nanograms (ng)/ milliliter (mL) | 0.940 (41.187) | 1.180 (39.076) | 1.750 (41.407) | 0.963 (47.672)
Statistical Analysis 1: Comparison: TV46046 Dose A vs Depo-subQ Provera; Test type: Other; Geometric Mean Ratio = 0.976, 90% CI 2-sided [0.748 to 1.274]
Statistical Analysis 2: Comparison: TV46046 Dose B vs Depo-subQ Provera; Test type: Other; Geometric Mean Ratio = 1.226, 90% CI 2-sided [0.940 to 1.598]
Statistical Analysis 3: Comparison: TV46046 Dose C vs Depo-subQ Provera; Test type: Other; Geometric Mean Ratio = 1.817, 90% CI 2-sided [1.380 to 2.392]

2. Primary Outcome: Time to Reach Cmax (Tmax) of MPA
Time Frame: Day 0 to Day 365
Population: PK analysis set included all randomized participants who received an injection of study drug, excluding any participants who had a baseline MPA concentration that exceeded 5% of their individual Cmax, had an important protocol deviation that may affect interpretation of their MPA data, or failed to provide at least 1 evaluable post-treatment MPA specimen.
Measure: Median (Full Range); unit: days
Arm/Group | TV46046 Dose A | TV46046 Dose B | TV46046 Dose C | Depo-subQ Provera
Number analyzed (Participants) | 16 | 15 | 14 | 14
days | 17.0 [1.0 to 105.0] | 28.0 [1.0 to 71.0] | 6.0 [2.0 to 336.0] | 31.5 [1.0 to 105.0]

3. Primary Outcome: Serum MPA Concentration at Day 91 (C91)
Time Frame: Day 91
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | TV46046 Dose A | TV46046 Dose B | TV46046 Dose C | Depo-subQ Provera
Number analyzed (Participants) | 16 | 15 | 14 | 14
ng/mL | 0.570 (36.802) | 0.660 (49.360) | 1.090 (40.151) | 0.474 (37.765)
Statistical Analysis 1: Comparison: TV46046 Dose A vs Depo-subQ Provera; Test type: Other; Geometric Mean Ratio = 1.202, 90% CI 2-sided [0.960 to 1.506]
Statistical Analysis 2: Comparison: TV46046 Dose B vs Depo-subQ Provera; Test type: Other; Geometric Mean Ratio = 1.393, 90% CI 2-sided [1.070 to 1.815]
Statistical Analysis 3: Comparison: TV46046 Dose C vs Depo-subQ Provera; Test type: Other; Geometric Mean Ratio = 2.301, 90% CI 2-sided [1.806 to 2.933]

4. Primary Outcome: Serum MPA Concentration at Day 182 (C182)
Time Frame: Day 182
Population: PK analysis set included all randomized participants who received an injection of study drug, excluding any participants who had a baseline MPA concentration that exceeded 5% of their individual Cmax, had an important protocol deviation that may affect interpretation of their MPA data, or failed to provide at least 1 evaluable post-treatment MPA specimen. Here, 'Overall number of participants analyzed' = participants evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | TV46046 Dose A | TV46046 Dose B | TV46046 Dose C | Depo-subQ Provera
Number analyzed (Participants) | 16 | 13 | 13 | 12
ng/mL | 0.201 (69.429) | 0.279 (65.793) | 0.443 (60.531) | 0.118 (150.789)
Statistical Analysis 1: Comparison: TV46046 Dose A vs Depo-subQ Provera; Test type: Other; Geometric Mean Ratio = 1.699, 90% CI 2-sided [0.921 to 3.135]
Statistical Analysis 2: Comparison: TV46046 Dose B vs Depo-subQ Provera; Test type: Other; Geometric Mean Ratio = 2.364, 90% CI 2-sided [1.273 to 4.390]
Statistical Analysis 3: Comparison: TV46046 Dose C vs Depo-subQ Provera; Test type: Other; Geometric Mean Ratio = 3.748, 90% CI 2-sided [2.033 to 6.908]

5. Primary Outcome: Serum MPA Concentration at Day 210 (C210)
Time Frame: Day 210
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | TV46046 Dose A | TV46046 Dose B | TV46046 Dose C | Depo-subQ Provera
Number analyzed (Participants) | 16 | 15 | 14 | 13
ng/mL | 0.119 (105.727) | 0.208 (76.683) | 0.365 (69.357) | 0.063 (244.107)
Statistical Analysis 1: Comparison: TV46046 Dose A vs Depo-subQ Provera; Test type: Other; Geometric Mean Ratio = 1.904, 90% CI 2-sided [0.886 to 4.093]
Statistical Analysis 2: Comparison: TV46046 Dose B vs Depo-subQ Provera; Test type: Other; Geometric Mean Ratio = 3.317, 90% CI 2-sided [1.585 to 6.942]
Statistical Analysis 3: Comparison: TV46046 Dose C vs Depo-subQ Provera; Test type: Other; Geometric Mean Ratio = 5.824, 90% CI 2-sided [2.796 to 12.135]

6. Primary Outcome: Area Under the Serum Drug Concentration-Time Curve From Time 0 to Day 182 (AUC0-182) of MPA
Time Frame: Day 0 to Day 182
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: days*ng/mL
Arm/Group | TV46046 Dose A | TV46046 Dose B | TV46046 Dose C | Depo-subQ Provera
Number analyzed (Participants) | 16 | 15 | 14 | 14
days*ng/mL | 94.2 (27.0) | 121.8 (38.1) | 173.6 (25.8) | 86.1 (29.6)
Statistical Analysis 1: Comparison: TV46046 Dose A vs Depo-subQ Provera; Test type: Other; Geometric Mean Ratio = 1.095, 90% CI 2-sided [0.920 to 1.302]
Statistical Analysis 2: Comparison: TV46046 Dose B vs Depo-subQ Provera; Test type: Other; Geometric Mean Ratio = 1.415, 90% CI 2-sided [1.148 to 1.744]
Statistical Analysis 3: Comparison: TV46046 Dose C vs Depo-subQ Provera; Test type: Other; Geometric Mean Ratio = 2.017, 90% CI 2-sided [1.692 to 2.405]

7. Primary Outcome: Area Under the Serum Drug Concentration-Time Curve From Time 0 to Day 210 (AUC0-210) of MPA
Time Frame: Day 0 to Day 210
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: days*ng/mL
Arm/Group | TV46046 Dose A | TV46046 Dose B | TV46046 Dose C | Depo-subQ Provera
Number analyzed (Participants) | 16 | 15 | 14 | 14
days*ng/mL | 100.2 (23.9) | 129.6 (37.8) | 187.0 (26.0) | 90.1 (27.6)
Statistical Analysis 1: Comparison: TV46046 Dose A vs Depo-subQ Provera; Test type: Other; Geometric Mean Ratio = 1.112, 90% CI 2-sided [0.948 to 1.303]
Statistical Analysis 2: Comparison: TV46046 Dose B vs Depo-subQ Provera; Test type: Other; Geometric Mean Ratio = 1.439, 90% CI 2-sided [1.174 to 1.762]
Statistical Analysis 3: Comparison: TV46046 Dose C vs Depo-subQ Provera; Test type: Other; Geometric Mean Ratio = 2.075, 90% CI 2-sided [1.751 to 2.459]

8. Primary Outcome: Area Under the Serum Drug Concentration-Time Curve From Time 0 to Infinity (AUC0-inf) of MPA
Time Frame: Day 0 to Day 365
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: days*ng/mL
Arm/Group | TV46046 Dose A | TV46046 Dose B | TV46046 Dose C | Depo-subQ Provera
Number analyzed (Participants) | 16 | 15 | 13 | 14
days*ng/mL | 117.2 (17.9) | 160.8 (36.6) | 224.9 (18.9) | 105.1 (19.5)
Statistical Analysis 1: Comparison: TV46046 Dose A vs Depo-subQ Provera; Test type: Other; Geometric Mean Ratio = 1.115, 90% CI 2-sided [0.993 to 1.252]
Statistical Analysis 2: Comparison: TV46046 Dose B vs Depo-subQ Provera; Test type: Other; Geometric Mean Ratio = 1.530, 90% CI 2-sided [1.277 to 1.833]
Statistical Analysis 3: Comparison: TV46046 Dose C vs Depo-subQ Provera; Test type: Other; Geometric Mean Ratio = 2.140, 90% CI 2-sided [1.888 to 2.425]

9. Primary Outcome: Apparent Terminal Half-life (t½) of MPA
Time Frame: Day 0 to Day 365
Population: as for outcome 4
Measure: Median (Full Range); unit: days
Arm/Group | TV46046 Dose A | TV46046 Dose B | TV46046 Dose C | Depo-subQ Provera
Number analyzed (Participants) | 16 | 15 | 13 | 14
days | 47.4 [18.7 to 114.8] | 85.3 [15.7 to 160.2] | 79.8 [19.4 to 130.4] | 37.4 [8.2 to 224.3]

10. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Time Frame: Day 0 up to Week 78
Population: Safety analysis set included all randomized participants who received an injection of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | TV46046 Dose A | TV46046 Dose B | TV46046 Dose C | Depo-subQ Provera
Number analyzed (Participants) | 16 | 15 | 14 | 15
Participants | 11 | 10 | 8 | 12

11. Secondary Outcome: Number of Participants With at Least 1 Concomitant Medication Use During Treatment
Description: Concomitant medications included acetic acid derivatives and substances, aminoalkyl ethers, anilides, calcium compounds, other viral vaccines, and propionic acid derivatives etc.
Time Frame: Day 0 up to Week 78
Population: Safety analysis set included all randomized participants who received an injection of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | TV46046 Dose A | TV46046 Dose B | TV46046 Dose C | Depo-subQ Provera
Number analyzed (Participants) | 16 | 15 | 14 | 15
Participants | 11 | 8 | 6 | 10

12. Secondary Outcome: Number of Participants With Clinically Significant Changes in Vital Signs
Description: Vital signs examination included blood pressure, respiration rate, pulse, and body temperature.
Time Frame: Day 0 to Day 365
Population: Safety analysis set included all randomized participants who received an injection of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | TV46046 Dose A | TV46046 Dose B | TV46046 Dose C | Depo-subQ Provera
Number analyzed (Participants) | 16 | 15 | 14 | 15
Participants | 0 | 0 | 0 | 0

13. Secondary Outcome: Change From Baseline in Body Weight at Day 7 and Weeks 13, 26, and 52
Time Frame: Day 7 and Weeks 13, 26, and 52
Population: Safety analysis set included all randomized participants who received an injection of study drug. Here, 'Number analyzed' = participants evaluable at specified timepoint.
Measure: Mean (Standard Error); unit: kilograms (kg)
Arm/Group | TV46046 Dose A | TV46046 Dose B | TV46046 Dose C | Depo-subQ Provera
Number analyzed (Participants) | 16 | 15 | 14 | 15
kilograms (kg)
  Change at Day 7 | -0.21 (0.19) | -0.27 (0.20) | -0.33 (0.17) | 0.05 (0.28)
  Change at Week 13 | -1.10 (1.42) | 0.92 (0.65) | 0.84 (0.35) | 1.40 (0.87)
  Change at Week 26: number analyzed (Participants) | 16 | 14 | 13 | 13
  Change at Week 26 | 1.14 (0.58) | 2.91 (1.11) | 1.38 (0.74) | 2.68 (0.89)
  Change at Week 52: number analyzed (Participants) | 16 | 13 | 14 | 14
  Change at Week 52 | 0.60 (0.56) | 1.38 (1.00) | 0.79 (1.06) | 1.99 (0.91)

14. Secondary Outcome: Number of Participants With Overall Opinion of Vaginal Bleeding Pattern
Description: Number of participants with overall opinion of vaginal bleeding pattern as acceptable or not acceptable has been reported.
Time Frame: Weeks 13, 26, and 52
Population: Safety analysis set included all randomized participants who received an injection of study drug. Here, 'Overall number of participants analyzed' = participants evaluable for this outcome measure. 'Number analyzed' = participants evaluable at specified timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | TV46046 Dose A | TV46046 Dose B | TV46046 Dose C | Depo-subQ Provera
Number analyzed (Participants) | 16 | 14 | 14 | 15
Participants
  Week 13: Acceptable | 10 | 9 | 11 | 11
  Week 13: Not Acceptable | 6 | 5 | 3 | 4
  Week 26: number analyzed (Participants) | 16 | 14 | 13 | 13
  Week 26: Acceptable | 12 | 13 | 9 | 12
  Week 26: Not Acceptable | 4 | 1 | 4 | 1
  Week 52: number analyzed (Participants) | 16 | 13 | 14 | 14
  Week 52: Acceptable | 14 | 12 | 13 | 13
  Week 52: Not Acceptable | 2 | 1 | 1 | 1

15. Secondary Outcome: Number of Participants With Patient Health Questionnaire (PHQ-9) Mood Scores
Description: The PHQ-9 is a participant-rated depressive symptom severity scale to monitor severity over time for newly diagnosed participants or participants in current treatment for depression. Scoring was based on participants' responses to each of the 9 questions, as follows: 0=not at all; 1=several days; 2=more than half the days; and 3=nearly every day. The PHQ-9 total score was calculated as the sum of the 9 individual item scores. The PHQ-9 total score was categorized as follows: 0 = no depression, 1 to 4=minimal depression, 5 to 9=mild depression, 10 to 14=moderate depression, 15 to 19=moderately severe depression; and 20 to 27=severe depression. Higher scores indicate more severe depression.
Time Frame: Baseline, Weeks 4, 13, 26, and 52
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | TV46046 Dose A | TV46046 Dose B | TV46046 Dose C | Depo-subQ Provera
Number analyzed (Participants) | 16 | 15 | 14 | 15
Participants
  Baseline: No Depression | 12 | 9 | 10 | 9
  Baseline: Minimal Depression | 4 | 4 | 3 | 5
  Baseline: Mild Depression | 0 | 2 | 1 | 1
  Baseline: Moderate Depression | 0 | 0 | 0 | 0
  Baseline: Moderately Severe Depression | 0 | 0 | 0 | 0
  Baseline: Severe Depression | 0 | 0 | 0 | 0
  Week 4: No Depression | 9 | 10 | 9 | 6
  Week 4: Minimal Depression | 5 | 4 | 3 | 7
  Week 4: Mild Depression | 1 | 1 | 1 | 1
  Week 4: Moderate Depression | 1 | 0 | 0 | 1
  Week 4: Moderately Severe Depression | 0 | 0 | 1 | 0
  Week 4: Severe Depression | 0 | 0 | 0 | 0
  Week 13: No Depression | 8 | 6 | 9 | 9
  Week 13: Minimal Depression | 6 | 7 | 5 | 4
  Week 13: Mild Depression | 2 | 2 | 0 | 1
  Week 13: Moderate Depression | 0 | 0 | 0 | 1
  Week 13: Moderately Severe Depression | 0 | 0 | 0 | 0
  Week 13: Severe Depression | 0 | 0 | 0 | 0
  Week 26: number analyzed (Participants) | 16 | 14 | 13 | 13
  Week 26: No Depression | 10 | 7 | 10 | 10
  Week 26: Minimal Depression | 4 | 5 | 2 | 2
  Week 26: Mild Depression | 2 | 2 | 1 | 1
  Week 26: Moderate Depression | 0 | 0 | 0 | 0
  Week 26: Moderately Severe Depression | 0 | 0 | 0 | 0
  Week 26: Severe Depression | 0 | 0 | 0 | 0
  Week 52: number analyzed (Participants) | 16 | 13 | 14 | 14
  Week 52: No Depression | 11 | 6 | 10 | 12
  Week 52: Minimal Depression | 4 | 5 | 3 | 2
  Week 52: Mild Depression | 1 | 1 | 0 | 0
  Week 52: Moderate Depression | 0 | 1 | 0 | 0
  Week 52: Moderately Severe Depression | 0 | 0 | 1 | 0
  Week 52: Severe Depression | 0 | 0 | 0 | 0

16. Secondary Outcome: Number of Participants With Clinically Significant Changes in Liver Function Tests
Time Frame: Day 0 to Day 365
Population: Safety analysis set included all randomized participants who received an injection of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | TV46046 Dose A | TV46046 Dose B | TV46046 Dose C | Depo-subQ Provera
Number analyzed (Participants) | 16 | 15 | 14 | 15
Participants | 0 | 0 | 0 | 0

17. Secondary Outcome: Estradiol Concentrations
Time Frame: Baseline, Weeks 4, 13, 26, 30, and 52
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: picograms (pg)/mL
Arm/Group | TV46046 Dose A | TV46046 Dose B | TV46046 Dose C | Depo-subQ Provera
Number analyzed (Participants) | 16 | 15 | 14 | 15
picograms (pg)/mL
  Baseline: number analyzed (Participants) | 16 | 15 | 13 | 15
  Baseline | 64.988 (57.169) | 52.825 (22.857) | 63.962 (74.815) | 66.181 (64.843)
  Week 4: number analyzed (Participants) | 16 | 15 | 14 | 14
  Week 4 | 72.357 (38.855) | 49.027 (48.373) | 31.149 (13.394) | 55.699 (28.077)
  Week 13 | 62.389 (56.316) | 45.890 (30.475) | 36.337 (25.065) | 42.071 (30.137)
  Week 26: number analyzed (Participants) | 16 | 13 | 13 | 13
  Week 26 | 114.347 (67.997) | 177.369 (197.661) | 52.132 (38.971) | 105.234 (67.421)
  Week 30: number analyzed (Participants) | 16 | 15 | 14 | 14
  Week 30 | 133.892 (138.964) | 77.861 (58.685) | 81.301 (58.232) | 142.691 (163.819)
  Week 52: number analyzed (Participants) | 16 | 13 | 14 | 14
  Week 52 | 122.994 (108.549) | 171.966 (166.209) | 148.441 (140.495) | 103.951 (63.290)

18. Secondary Outcome: Number of Participants With No Ovulation in 12 Months
Description: Ovulation was defined as one or more progesterone measurements ≥ 4.7 ng/mL in Weeks 48, 49, 50, 51 or 52.
Time Frame: 12 months
Population: Safety analysis set included all randomized participants who received an injection of study drug. Here, 'Overall number of participants analyzed' = participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | TV46046 Dose A | TV46046 Dose B | TV46046 Dose C | Depo-subQ Provera
Number analyzed (Participants) | 15 | 13 | 13 | 13
Participants | 4 | 7 | 8 | 3

19. Secondary Outcome: Number of Participants With 1 or More Injection Site Reactions (ISRs)
Description: The ISRs included erythema, swelling, pruritus, bleeding, tenderness, bruising, hypopigmentation, atrophy, and injection site pain.
Time Frame: Day 0 to Day 365
Population: Safety analysis set included all randomized participants who received an injection of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | TV46046 Dose A | TV46046 Dose B | TV46046 Dose C | Depo-subQ Provera
Number analyzed (Participants) | 16 | 15 | 14 | 15
Participants | 7 | 6 | 6 | 4

20. Secondary Outcome: Number of Participants With Responses to the Acceptability Question (What do You Like About the Method?)
Description: Acceptability questions include likes and dislikes of the method and willingness to use the product in the future.
Time Frame: Weeks 26 and 52
Population: Safety analysis set included all randomized participants who received an injection of study drug. Here, 'Overall number of participants analyzed' = participants evaluable for this outcome measure. 'Number analyzed' = participants evaluable for specified category.
Measure: Count of Participants; unit: Participants
Arm/Group | TV46046 Dose A | TV46046 Dose B | TV46046 Dose C | Depo-subQ Provera
Number analyzed (Participants) | 16 | 13 | 14 | 14
Participants
  Week 26: Easy to use: number analyzed (Participants) | 16 | 12 | 13 | 13
  Week 26: Easy to use | 7 | 7 | 7 | 8
  Week 26: Weight gain: number analyzed (Participants) | 16 | 12 | 13 | 13
  Week 26: Weight gain | 2 | 1 | 4 | 1
  Week 26: Weight loss: number analyzed (Participants) | 16 | 12 | 13 | 13
  Week 26: Weight loss | 1 | 1 | 0 | 0
  Week 26: Menstrual changes: number analyzed (Participants) | 16 | 12 | 13 | 13
  Week 26: Menstrual changes | 6 | 5 | 3 | 5
  Week 26: Discreet: number analyzed (Participants) | 16 | 12 | 13 | 13
  Week 26: Discreet | 8 | 8 | 4 | 5
  Week 26: Provides longer-term protection than other method: number analyzed (Participants) | 16 | 12 | 13 | 13
  Week 26: Provides longer-term protection than other method | 6 | 4 | 4 | 3
  Week 26: Few side effects: number analyzed (Participants) | 16 | 12 | 13 | 13
  Week 26: Few side effects | 5 | 5 | 6 | 2
  Week 26: Has to be administered by a healthcare provider: number analyzed (Participants) | 16 | 12 | 13 | 13
  Week 26: Has to be administered by a healthcare provider | 2 | 3 | 2 | 3
  Week 26: Nothing: number analyzed (Participants) | 16 | 12 | 13 | 13
  Week 26: Nothing | 1 | 0 | 0 | 0
  Week 26: Other: number analyzed (Participants) | 16 | 12 | 13 | 13
  Week 26: Other | 1 | 1 | 0 | 1
  Week 52: Easy to use | 13 | 11 | 10 | 11
  Week 52: Weight gain | 2 | 4 | 3 | 1
  Week 52: Weight loss | 2 | 1 | 0 | 0
  Week 52: Menstrual changes | 5 | 4 | 3 | 4
  Week 52: Discreet | 7 | 6 | 6 | 9
  Week 52: Provides longer-term protection than other method | 7 | 8 | 3 | 10
  Week 52: Few side effects | 10 | 5 | 7 | 6
  Week 52: Has to be administered by a healthcare provider | 2 | 2 | 1 | 2
  Week 52: Nothing | 0 | 1 | 0 | 0
  Week 52: Other | 0 | 0 | 0 | 0

21. Secondary Outcome: Number of Participants With Responses to the Acceptability Question (What do You Not Like About the Method?)
Description: Acceptability questions include likes and dislikes of the method and willingness to use the product in the future.
Time Frame: Weeks 26 and 52
Population: as for outcome 20
Measure: Count of Participants; unit: Participants
Arm/Group | TV46046 Dose A | TV46046 Dose B | TV46046 Dose C | Depo-subQ Provera
Number analyzed (Participants) | 16 | 13 | 14 | 14
Participants
  Week 26: Pain at injection: number analyzed (Participants) | 16 | 12 | 13 | 13
  Week 26: Pain at injection | 2 | 1 | 3 | 1
  Week 26: Once injected, it cannot be reversed: number analyzed (Participants) | 16 | 12 | 13 | 13
  Week 26: Once injected, it cannot be reversed | 2 | 1 | 0 | 0
  Week 26: Weight gain: number analyzed (Participants) | 16 | 12 | 13 | 13
  Week 26: Weight gain | 1 | 6 | 5 | 6
  Week 26: Weight loss: number analyzed (Participants) | 16 | 12 | 13 | 13
  Week 26: Weight loss | 0 | 0 | 0 | 0
  Week 26: Nothing: number analyzed (Participants) | 16 | 12 | 13 | 13
  Week 26: Nothing | 5 | 2 | 2 | 5
  Week 26: Menstrual changes: number analyzed (Participants) | 16 | 12 | 13 | 13
  Week 26: Menstrual changes | 7 | 6 | 8 | 4
  Week 26: Injection site reactions: number analyzed (Participants) | 16 | 12 | 13 | 13
  Week 26: Injection site reactions | 0 | 0 | 0 | 0
  Week 26: Other side effects: number analyzed (Participants) | 16 | 12 | 13 | 13
  Week 26: Other side effects | 3 | 0 | 0 | 1
  Week 26: Other: number analyzed (Participants) | 16 | 12 | 13 | 13
  Week 26: Other | 0 | 0 | 0 | 1
  Week 52: Pain at injection | 2 | 2 | 2 | 1
  Week 52: Once injected, it cannot be reversed | 4 | 3 | 0 | 0
  Week 52: Weight gain | 1 | 4 | 6 | 6
  Week 52: Weight loss | 1 | 0 | 0 | 0
  Week 52: Nothing | 5 | 1 | 3 | 5
  Week 52: Menstrual changes | 8 | 8 | 6 | 3
  Week 52: Injection site reactions | 1 | 2 | 1 | 0
  Week 52: Other side effects | 1 | 2 | 0 | 1
  Week 52: Other | 0 | 0 | 0 | 0

22. Secondary Outcome: Number of Participants With Responses to the Acceptability Question (If You Were at Risk for Pregnancy, Would You Use This Method of Contraception Outside of This Study?)
Description: Acceptability questions include likes and dislikes of the method and willingness to use the product in the future.
Time Frame: Weeks 26 and 52
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | TV46046 Dose A | TV46046 Dose B | TV46046 Dose C | Depo-subQ Provera
Number analyzed (Participants) | 16 | 12 | 14 | 14
Participants
  Week 26: number analyzed (Participants) | 15 | 12 | 12 | 12
  Week 26: Yes | 4 | 2 | 2 | 3
  Week 26: No | 11 | 10 | 10 | 9
  Week 52: Yes | 2 | 2 | 3 | 2
  Week 52: No | 14 | 10 | 11 | 12

23. Secondary Outcome: Number of Participants With Responses to the Acceptability Question (If You Had a Choice, Which Injectable Contraceptive Method Would You Prefer?)
Description: Acceptability questions include likes and dislikes of the method and willingness to use the product in the future.
Time Frame: Weeks 26 and 52
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | TV46046 Dose A | TV46046 Dose B | TV46046 Dose C | Depo-subQ Provera
Number analyzed (Participants) | 16 | 13 | 13 | 14
Participants
  Week 26: number analyzed (Participants) | 16 | 12 | 13 | 13
  Week 26: Injection every 1 month | 0 | 1 | 0 | 0
  Week 26: Injection every 3 months | 3 | 3 | 3 | 2
  Week 26: Injection every 6 months | 6 | 5 | 5 | 4
  Week 26: Injection every 12 months | 5 | 3 | 5 | 5
  Week 26: Frequency of reinjections is not important | 2 | 0 | 0 | 2
  Week 52: Injection every 1 month | 0 | 0 | 0 | 0
  Week 52: Injection every 3 months | 3 | 2 | 2 | 1
  Week 52: Injection every 6 months | 2 | 4 | 3 | 5
  Week 52: Injection every 12 months | 10 | 6 | 7 | 6
  Week 52: Frequency of reinjections is not important | 1 | 1 | 1 | 2

24. Secondary Outcome: Progesterone Concentration
Time Frame: Weeks 48, 49, 50, 51, and 52
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | TV46046 Dose A | TV46046 Dose B | TV46046 Dose C | Depo-subQ Provera
Number analyzed (Participants) | 16 | 13 | 14 | 14
ng/mL
  Week 48: number analyzed (Participants) | 15 | 13 | 12 | 14
  Week 48 | 2.103 (3.993) | 0.945 (2.422) | 2.255 (4.395) | 2.682 (3.900)
  Week 49: number analyzed (Participants) | 16 | 13 | 14 | 13
  Week 49 | 1.803 (3.268) | 2.448 (3.784) | 1.593 (3.471) | 4.323 (5.276)
  Week 50: number analyzed (Participants) | 16 | 13 | 14 | 13
  Week 50 | 4.793 (6.791) | 5.224 (7.554) | 1.649 (3.085) | 3.086 (5.312)
  Week 51: number analyzed (Participants) | 16 | 12 | 14 | 13
  Week 51 | 4.280 (7.133) | 0.795 (0.928) | 1.214 (2.737) | 1.669 (3.390)
  Week 52 | 2.096 (4.319) | 2.264 (4.167) | 2.561 (5.069) | 2.529 (4.152)

ADVERSE EVENTS:
Time Frame: Day 0 up to Week 78
Description: Safety analysis set included all randomized participants who received an injection of study drug.
Arm/Group | TV46046 Dose A | TV46046 Dose B | TV46046 Dose C | Depo-subQ Provera
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/15 | 0/14 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/15 | 0/14 | 1/15
Other Adverse Events (participants affected / at risk) | 11/16 | 10/15 | 8/14 | 12/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TV46046 Dose A (N=16) | TV46046 Dose B (N=15) | TV46046 Dose C (N=14) | Depo-subQ Provera (N=15)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TV46046 Dose A (N=16) | TV46046 Dose B (N=15) | TV46046 Dose C (N=14) | Depo-subQ Provera (N=15)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (3)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 2 (2) | 2 (2) | 1 (1) | 1 (1)
Injection site erythema (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Injection site pain (General disorders) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acarodermatitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Amoebic dysentery (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bacterial vaginosis (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Bronchitis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Furuncle (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mastitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Tinea infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Vulvovaginal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Postoperative ileus (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Weight increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Increased appetite (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 6 (8) | 2 (4) | 1 (1) | 4 (4)
Sinus headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Adjustment disorder with depressed mood (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (2) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Metrorrhagia (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Nipple pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Reflux laryngitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hidradenitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.

DOCUMENTS (2):
  • Study Protocol (2021-03-16): https://cdn.clinicaltrials.gov/large-docs/53/NCT04682353/Prot_000.pdf
  • Statistical Analysis Plan (2023-02-15): https://cdn.clinicaltrials.gov/large-docs/53/NCT04682353/SAP_001.pdf